CLINICAL TRIAL: NCT02391753
Title: Optimal Time For Evaluation of Labor Related Pelvic Floor Changes: A 3D Transperineal Ultrasound Study
Brief Title: Evaluation of Labor Related Pelvic Floor Changes: A 3D Transperineal Ultrasound Study
Acronym: OTELaPFC
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: BVU1/13-1
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Pelvic Floor Disorders
Keywords: levator avulsion; transperineal ultrasound; levator hiatus
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Transperineal 3D Ultrasound — Imaging was performed with women in lithotomy position with empty bladder. The probe was covered with a sterile film and placed on the perineum in the sagittal plane. The field of view angle was set to a maximum of 70° in the sagittal plane and the volume acquisition angle to 85° in the axial plane. Analysis of stored volumes was conducted offline by another experienced investigator blinded to clinical and delivery data.

SUMMARY:
The aim of the study was the define changes LAM morphology, biometric measurements of the LAM and genital hiatus at immediate evaluation of pelvic floor and at 3 month after delivery was evaluated. We also sought to define the optimal time for evaluation of pelvic floor after childbirth

DETAILED DESCRIPTION:
Sixty four of 72 primiparous women who vaginally delivered singleton babies that eligible for trial were examined within 36 h of delivery and at 3rd months after delivery.Parameters such as age, episiotomy, mode of delivery, duration of labor, birthweight and antenatal biparietal diameter (BPD) measures were obtained from the clinical files. The length of the first stage of labor was calculated from the beginning of regular and at least three strong uterine contractions in 30 min according to the women's statements, tocography and palpations to full dilatation. All static ultrasound volume acquisitions were performed by the same experienced sonographer trained in pelvic floor ultrasound within 36 h of delivery. Same patients invited for second evaluation.Two 3-D volumes (one at rest, one on Valsalva maneuver) were recorded in the supine position after voiding.The effectiveness of valsalva was ascertained by observing 2-D ultrasounds before acquiring volumes.. LAM thickness is determined at the plane of minimal hiatal dimensions rather than 1-1.5 cm above the actual LAM hiatus where LAM thickness is maximal as described by Dietz et al.(15). The following parameters were assessed for this study: maximum diameters of the LAM hiatus (anteroposterior and transverse) at rest and on Valsalva maneuver; area of the LAM hiatus at rest and on Valsalva; and pubovisceral muscle thickness (left and right of the rectum), difference in anteroposterior and transverse diameter of hiatus and LAM hiatus area between rest and Valsalva

ELIGIBILITY:
Inclusion Criteria:

* primiparous women who vaginally delivered singleton babies that eligible for trial were examined within 36 h of delivery

Exclusion Criteria:

* operative deliveries (forceps or vacuum assisted), multifetal pregnancy, cesarean delivery, handicap in lithotomy position, refused consent and uncooperative patient for effective Valsalva maneuver.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: primiparous women who vaginally delivered singleton babies that eligible for trial were examined within 36 h of delivery
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Levator Avulsion | 01.07.2014